CLINICAL TRIAL: NCT06663735
Title: A Cross-sectional Study Describing the Current Status of Diagnosis and Treatment of Uroepithelial Cancer in Hospitals of Different Grades in Henan Province
Brief Title: Current Status of Diagnosis and Treatment of Uroepithelial Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: CHASE010
Record Dates: First submitted 2024-10-21; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Uroepithelial Carcinoma
Keywords: Henan province; uroepithelial cancer; treatment
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 400 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnosis and management of patients with early stage resectable uroepithelial carcinoma: The study is a multicenter, non-interventional, observational cross-sectional study. It is planned to enroll patients with early stage resectable uroepithelial cancer in each study hospital in Henan Province. This is a cross-sectional study, and all patients will be anonymized for clinical data collection, and detailed information on patient demographic characteristics as well as medical and treatment history, hospitals at different stages of treatment, pathological test results, and medication regimens will be recorded at the beginning of enrollment.
- Diagnosis and management of patients with advanced unresectable uroepithelial cancer: It is planned to enroll patients with advanced unresectable uroepithelial cancer in each study hospital in Henan Province. This is a cross-sectional study, and all patients will be anonymized for clinical data collection, and detailed information on patient demographic characteristics as well as medical and treatment history, hospitals at different stages of treatment, pathological test results, and medication regimens will be recorded at the beginning of enrollment.

SUMMARY:
A cross-sectional study describing the current status of diagnosis and treatment of uroepithelial cancer in hospitals of different grades in Henan Province

DETAILED DESCRIPTION:
Patients diagnosed with uroepithelial carcinoma attending multiple research center hospitals in Henan Province from January 1, 2023 to December 31, 2023 A questionnaire was used to collect and analyze the treatment patterns of patients with early versus advanced uroepithelial cancer in different levels of hospitals in Henan Province.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age (at enrollment)
* Histologically confirmed uroepithelial carcinoma
* Patients with newly diagnosed or completed radical uroepithelial carcinoma in the early stages of uroepithelial cancer/advanced unresectable or with distant metastases of urothelial carcinoma
* Complete medical history information

Exclusion Criteria:

* Incomplete medical history and medical records

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with uroepithelial carcinoma attending multiple research center hospitals in Henan Province from January 1, 2023-December 31, 2023
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Describing the diagnosis and treatment patterns of patients with early versus advanced uroepithelial carcinoma in different grades of hospitals in Henan Province | up to the patients enrolled,an average of 1 year
  To describe the similarities and differences between the way patients with early and advanced uroepithelial cancer are diagnosed and treated in different levels of hospitals in Henan Province and the current guidelines for uroepithelial cancer.

SECONDARY OUTCOMES:
Comparison of differences in diagnosis and treatment patterns between patients with early-stage and advanced uroepithelial carcinoma in county hospitals and different consultation departments of the same hospital in Henan province | up to the patients enrolled,an average of 1 year
  The main purpose of this study is to compare the differences between the diagnosis and treatment modalities and guidelines for early and advanced uroepithelial cancer patients in Henan Province in county hospitals. It also compares the differences in treatment modalities between different departments in the same level of hospitals.
Describing the pathology as well as genetic testing of patients with uroepithelial carcinoma in different grades of hospitals in Henan province | up to the patients enrolled,an average of 1 year
  1. Proportion of different genes/proteins tested in patients with uroepithelial cancer (mutations in FGFR, HER2, HRR, ARID1A and CREBBP, TP53, CDKN2A and PD-L1 expression)
  2. Proportion of early and advanced uroepithelial cancer patients with high expression/mutations of different genes and use of targeted therapies

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Kaifeng City Center Hospital, Kaifeng, Henan
  - Luoyang Renda Hospital, Luoyang, Henan
  - Nanyang City Center Hospital, Nanyang, Henan
  - Qingfeng County People's Hospital, Puyang, Henan
  - Department of Oncology, Xinxiang, Henan
  - Hui County People's Hospital, Xinxiang, Henan
  - Jun County People's Hospital, Xinxiang, Henan
  - Qi County People's Hospital, Xinxiang, Henan
  - Xinxiang Allied Hospital, Xinxiang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No